CLINICAL TRIAL: NCT06332469
Title: Feasibility Study of an Internet Based Education and Support Program for Patients Awaiting Kidney Transplantation
Brief Title: Evaluation of an Internet Based Education and Support Program for Patients Awaiting Kidney Transplantation
Acronym: INSERT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Kristina Nilsson, MSc, PhD-student, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INSERT feasibility
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
Keywords: kidney transplantation; psychosocial support; patient education; e-health
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The intervention group gets immediate access to the 9 week program, and the waitlist control group gets access after a 9 week waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): This group gets immediate access to the program
  Interventions: Behavioral: Internet based education and support program for patients awaiting kidney transplantation
- Wailtlist group (No Intervention): This group gets access to the same program after a 9 week waiting time

INTERVENTIONS:
Behavioral: Internet based education and support program for patients awaiting kidney transplantation — A guided internet based support an education program consisting of 9 modules running over 9 weeks. First, an introductory module is given that involves goal setting, followed by two educational modules with information regarding kidney disease, treatment and self-care in severe renal failure and while waiting for kidney transplantation, and kidney transplant-specific areas. Supportive content consist of three behavioral components spread over five modules/weeks and are based on cognitive behavioural therapy principles. The last module is a summation focusing on consolidating the knowledge learned during the program.
  Each module consists of texts, illustrations, short films, reminders to practice physical activity and weekly homework for which the participants receive feedback from a contact person.
  Arms: Treatment group

SUMMARY:
The goal of this study is to test the feasibility study of an internet based education and support program for patients awaiting kidney transplantation. The study is designed as a national pilot randomized controlled trial with a waitlist control group, to test the feasibility, acceptability, and potential effects of the intervention on patients' physical and mental health.

DETAILED DESCRIPTION:
Persons 18 years and older with severe renal failure and accepted on waiting list for kidney transplant with deceased donor in Sweden since at least 6 months will be recruited for participation.

Recruitment will be performed through Sweden's four transplant centers. Exclusion criteria will include not considering themselves able to spend 3-4 hours/week to work in the program. The study will be performed using a study platform which is previously well tested.

The intervention group The intervention is a support an education program, consisting of 9 modules running over 9 weeks. First, an introductory module is given that involves goal setting, followed by two training modules with information; The first on kidney disease, treatment and self-care in severe renal failure and while waiting for kidney transplantation, the second on kidney transplant-specific areas such as drugs, potential complications, lifestyle advice and self-care before and after kidney transplantation. This is followed by three behavioral components spread over five modules/weeks: acceptance (one module), problem solving (one module) and behavioral activation (three modules), and finally a summation module that focuses on consolidating the knowledge learned during the program. Each module consists of texts, illustrations, short films, reminders to practice physical activity and weekly homework for which the people receive feedback from a contact person. Any participants who are transplanted while undergoing the program will be offered to continue the study with adapted modules. Adaptations involve more relevant examples and information regarding drugs, complications and diet which become more relevant after the transplant.

Waitlist control group The control group will be followed with weekly check-ups for 9 weeks via the study platform regarding well-being, whether they have been transplanted or if something happened that affects their life situation. After the intervention period of 9 weeks, the control group will be offered the same program as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* severe renal failure and accepted on waiting list for kidney transplant with deceased donor in Sweden since at least 6 months

Exclusion Criteria:

* Not considering themselves able to spend 3-4 hours/week to work in the program
* Another illness that permanently renders kidney transplantation impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Kidney transplant understanding tool (K-TUT) | 9 weeks
  The Kidney Transplant Understanding Tool (K-TUT) is an instrument to assess patient knowledge about kidney transplantation, consisting of 9 true and false, and 13 multiple-choice questions (each with more than 1 potential answer). In total, 69 items address several aspects related to kidney transplantation. Each statement is dichotomized ("correct" or "incorrect"). One point is given for each correct answer chosen, and the scores are summed and converted to percentages. A perfect score (100%) equates to a total of 69 points.
Self-care in chronic illness inventory v.4c | 9 weeks
  A self-report instrument with four scales; the self-care maintenance scale has 7 items, the self-care monitoring scale has 5 items, the self-care management scale has 6 items, and lastly the self-care confidence scale has 10 items. The latter was added after studies showed that self-efficacy is a major predictor of self-care. Each SC-CII item is measured using a 5-point likert scale ranging from "Never" (1) to "Always" (5), "Not likely" (1) to "Very likely" (5) and "Not confident" (1) to "Very confident" (5). The scales use a standardized score from 0 to 100, with higher scores indicating better self-care.
The Self-Efficacy for Managing Chronic Disease 6-item Scale (SES6G | 9 weeks
  The Self-Efficacy for Managing Chronic Disease 6-item Scale (SES6G) is a tool designed to assess an individual's confidence in their ability to manage the various aspects of living with a chronic illness. It is a short form of the original Self-Efficacy for Managing Chronic Disease 8-item Scale (SES8G). The scoring involves participants rating their confidence on a numerical scale (e.g., from 1 to 10) for each item. The scores are summed to obtain a total score. Higher scores indicate greater self-efficacy in managing chronic disease, reflecting a higher level of confidence in one's ability to handle the challenges associated with the condition.
Pearlin Mastery Scale | 9 weeks
  The Pearlin Mastery Scale is a self-report instrument designed to measure the extent to which individuals perceive control over their lives and events that affect them. It assesses the concept of "psychological mastery," which refers to an individual's perceived ability to control and influence outcomes in their life.
  The Pearlin Mastery Scale consists of 7 items where respondents are asked to rate their level of agreement or disagreement with each statement, reflecting their perceived mastery or control. The scale is scored by summing the responses to the individual items, providing an overall score that indicates the level of perceived mastery. Higher scores suggest a greater sense of mastery or perceived control, while lower scores may indicate a lower sense of control. Response options consist of a Likert scale which ranges from 1, strongly disagree to 4, strongly agree [4-point]. The items are summed, with higher scores indicating greater mastery/self-efficacy.
The Depression Anxiety Stress Scales 21 (DASS-21) | the last week
  The Depression Anxiety Stress Scales 21 (DASS-21) is a self-report instrument designed to measure and assess levels of depression, anxiety, and stress in individuals. It is a shortened version of the DASS-42, consisting of 21 questions. The DASS-21 is intended to provide a quick and efficient overview of an individual's mental health.
  The scoring for the Depression Anxiety Stress Scales 21 (DASS-21) involves calculating separate scores for each of the three subscales: Depression, Anxiety and Stress. Each subscale contains seven items, and participants rate the extent to which they have experienced each symptom over the past week on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). DASS-21 provides separate scores for each subscale, where higher scores on each subscale indicate higher levels of depression, anxiety or stress.
Acceptance of chronic health conditions scale (ACHC) | 9 weeks
  The Acceptance of Chronic Health Conditions (ACHC) Scale is a self-report measure of acceptance in chronic health conditions. The ACHC Scale consists of 10 items scored on a 5-category Likert rating scale. Four items are positively worded, and 6 negatively worded. The ratings are summed; in the summation of the score the positively worded items are coded in reverse. A high total sum score indicates a high level of acceptance, and a low sum score indicates a low level of acceptance.
EQ-5D-5L | 9 weeks
  A self-report instrument measuring health related quality of life, with one question for each of the five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Marking a level results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The instrument also has a visual analogue scale where 'The best health you can image' (=100) and 'The worst health you can image' (=0). This scale can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Nilsson, MSc, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Linköping University,, Norrköping
  - Linköping University, Norrköping

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data as this is considered sensitive information

REFERENCES:
- [Background] Nilsson K, Westas M, Andersson G, Johansson P, Lundgren J. Waiting for kidney transplantation from deceased donors: Experiences and support needs during the waiting time -A qualitative study. Patient Educ Couns. 2022 Jul;105(7):2422-2428. doi: 10.1016/j.pec.2022.02.016. Epub 2022 Feb 22. PMID 35272905
- [Background] Nilsson K, Andersson G, Johansson P, Lundgren J. Developing and designing an internet-based support and education program for patients awaiting kidney transplantation with deceased donors through: a Delphi study. BMC Nephrol. 2023 Oct 25;24(1):311. doi: 10.1186/s12882-023-03364-2. PMID 37880582
- See also: The study web platform where study information is available and potential participants can register their interest of participation. — http://www.iterapi.se/sites/insert/